# UPMC CancerCenter

Partner with University of Pittsburgh Cancer Institute

**Title**: A Phase II Prospective Trial of Low-Level Laser Therapy for Prevention of Oral Mucositis in Patients Receiving Chemotherapy and Radiation for Head and Neck Cancer

Version: 12/03/2015

## **Principal Investigator:**

David A. Clump, MD, PhD Assistant Professor Department of Radiation Oncology University of Pittsburgh Cancer Institute 5230 Centre Avenue Pittsburgh, PA 15232 clumpda2@upmc.edu Ph. (412) 623-6720 Fax (412) 623-6192

## **Co-investigators:**

Dwight Heron, MD Brian Karlovits, DO Julie Bauman, MD James Ohr, DO

#### Statistician:

Hong Wang, PhD

# **Table of Contents**

| Study | y Schema | 4 |
|---|---|---|
| 1.0<br>1.1<br>1.2 | · / - · | 5 |
| 2.1<br>2.2<br>2.3<br>2.4 | Product Background Product Mechanism of Action Product Efficacy Table 1. LLLT trials for oral mucositis prevention Product Safety | |
| 3.0<br>3.1<br>3.2<br>3.3 | Patient Selection | 9<br>10 |
| <b>4.1</b> | 4.1.1 Definition of Target Volumes: 4.1.2 Definition of Organs at Risk: Chemotherapy Low-Level Laser Therapy | 1111111112 |
| 5.0<br>5.1<br>5.2 | | 13 |
| 6.0<br>6.1<br>6.2<br>6.3<br>6.4<br>6.5<br>6.6<br>6.7<br>6.8<br>6.9 | Secondary Endpoints: Exploratory Endpoints: Sample Size | |
| 7.0<br>7.1<br>7.2<br>7.3<br>7.4<br>7.5 | Adverse Event Characteristics | |
| 8.0 | Registration Procedures | 23 |

| 8.2 | Registration Process | 23 |
|------|---------------------------------------------------------|----|
| 9.0 | Protocol Conduct and Guidelines | 24 |
| 9.1 | Protocol amendments, or changes in study conduct | 24 |
| | Publication of results | |
| 9.3 | Ethics and Good Clinical Practice | 24 |
| 9.4 | Institutional Review Board/Independent Ethics Committee | 24 |
| | Informed consent | |
| 9.6 | Declaration of Helsinki | 25 |
| 10.0 | References | 26 |

# **Study Schema**

A phase II, single-arm trial to examine the efficacy of prophylactic low-level laser therapy (LLLT) to reduce the incidence of oral mucositis and adverse events in patients receiving combined modality therapy consisting of chemotherapy and radiation therapy for head and neck cancer.

Patients meeting the eligibility criteria will be enrolled to receive prophylactic LLLT in addition to standard of care measures for oral mucositis or other toxicity of therapy. The radiation and chemotherapy dose, schedule, modality, technique, and any required adjustments will not be influenced by this protocol and will follow standard existing institutional practices.

Patients will receive LLLT three times per week concurrently with chemoradiotherapy. LLLT may be delivered either immediately prior to or after the patient's daily fraction of radiotherapy. Patients will be treated extra-orally with a THOR® LED cluster for one minute along the buccal mucosa on each side and intraorally for one minute to the tongue and soft palate. During each LLLT treatment session a thorough oral exam will be performed to identify any areas of mucositis. If the patient should develop intraoral lesions they will be targeted directly with the intraoral probe for one minute to each site of mucositis. The laser settings to be used are as follows: frequency 2.5 Hz; wavelength 660 nm; and power 75 mW, for an energy of 4.5 J.

Patients will be evaluated prior to therapy, weekly during therapy, two weeks after the completion of therapy, and three months after the completion of therapy. During each assessment, the following toxicities will be assessed: pain, mucositis, dysphagia, xerostomia, dysgeusia, dermatitis, trismus, and quality of life.

Previous studies indicate that approximately 40% of patients will experience severe mucositis with radiation and concurrent chemotherapy. The hypothesis in this trial is that the addition of LLLT to this treatment regimen will decrease the rate of severe acute OM to 20%. We plan to enroll 50 patients at our institution in 12 months after the trial opens.

# 1.0 Objectives:

### 1.1 Primary Objective

Our primary objective is to determine the ability of low-level laser therapy (LLLT) to reduce the rates of severe oral mucositis in patients receiving radiation with concurrent chemotherapy for head and neck cancer (HNC).

## 1.2 Secondary Objectives

- 1. To establish the time to onset of severe oral mucositis following the initiation of radiotherapy with LLLT.
- 2. To determine the incidence of pain, dysphagia, xerostomia, dysgeusia, trismus, radiodermatitis, and OM-related QOL (via FACT-H&N score) with LLLT.
- 3. To evaluate the mean cumulative radiation dose at time of onset of severe oral mucositis with LLLT.
- 4. Determine the duration of oral mucositis.
- 5. Record the amount of narcotic analgesia use during treatment.
- 6. Evaluate the number of breaks in chemoradiotherapy with LLLT use.
- 7. Determine the proportion of patients who require feeding tube placement during treatment.

### 2.0 Introduction

### 2.1 Disease Overview

Combined modality therapy with chemotherapy and radiation is a commonly employed treatment approach for patients with various types of HNC [1]. Despite the overall safety and efficacy of this treatment modality, side effects exist, including acute chemoradiation-induced pain, dermatitis, xerostomia, dysgeusia, dysphagia, odynophagia, and oral mucositis. In fact, a majority of patients treated with this modality will experience some degree of oral mucositis (OM) [2]. OM can affect many oral functions including mastication and swallowing which may lead to dehydration, renal failure and necessitate the placement and use of a feeding tube and negatively impact and patient's quality of life (QOL). Severe OM can also predispose a patient to increased risk of infections requiring hospitalization and increased cost of treatment [3]. The severity of these reactions can be so severe that patients who experience treatment-related mucositis are less likely to complete the planned course of therapy without unplanned interruptions in therapy. Previous studies provide evidence that unplanned breaks in radiotherapy for HNC result in worse tumor control [4]. Furthermore, adverse events can increase the cost of healthcare by resulting in preventable hospital admissions for intravenous hydration and nutritional support and procedures including feeding tube placement. In fact, OM has been shown to be associated with an incremental cost of \$1,700 - \$6,000 per patient, depending on the grade [5].

Despite multiple clinical trials, no single treatment has been proven to be effective in substantially reducing incidence or severity of chemoradiation induced oral mucositis. The current standard practice for the management of OM is symptom management and supportive care with narcotic pain medications and anesthetic mouth rinses and nutritional support with supplementation either by mouth or feeding tube.

### 2.2 Product Background

Photomedicine utilizing low level laser (or "light" as light emitting diode sources are increasingly being used in place of lasers) therapy (LLLT) has been investigated as a novel therapeutic approach since the 1960s. LLLT is a safe, low-intensity form of light therapy. LLLT employs visible (generally red) or near-infrared light generated from a laser or light emitting diode (LED) [6]. Therapy with LLLT has been shown to relieve pain, reduce inflammation, and improve tissue repair. LLLT does not function through ablative or thermal mechanisms, but rather a photochemical effect comparable to photosynthesis in plants whereby the light is absorbed and exerts a chemical change [6].

LLLT was first completely limited to treatment with laser sources, such as the helium neon (HeNe) or indium phosphide, gallium and aluminum diode (InGaAIP) lasers. The non-coherent light produced by light emitting diode (LED) devices has the same biological properties and clinical effectiveness as coherent light produced by lasers, with the advantages of LED technology being that it is significantly less expensive and can be arranged in arrays permitting greater surface area exposure and subsequent shorter overall treatment times. Furthermore, LED-based LLLT applied extraorally has good penetration through skin and soft tissue to the oral mucosa [7]

#### 2.3 Product Mechanism of Action

The mechanism of action no LLLT is rooted in photochemistrisy. Light photons must be absorbed by molecular photoacceptors or chromophores for photochemistry to occur [8]. The cellular mechanism of LLLT has been attributed to the absorption of monochromatic visible and near infrared (NIR) radiation by the cellular respiratory chain [9]. Phototherapy is characterized by its ability to induce photobiological processes in cells. Mitochondria play a crucial role in cellular metabolism and the generation of energy in the form of adenosine triphosphate (ATP) through oxidative phosphorylation. Mitochondria have been studied as the main target of phototherapy. Cytochrome c oxidase is the proposed photoacceptor for the red-NIR light range in mammalian cells, as absorption spectra for light were found to be similar to the absorption spectra of cytochrome c oxidase [10]. LLLT to isolated mitochondria increased ATP synthesis, RNA and protein synthesis, and enhanced synthesis of NADH and ATP [6]. In stressed tissues, mitochondria make nitric oxide that competes with oxygen in the oxidative phosphorylation chain. This in turn decreases ATP synthesis and can increase production

of reactive oxygen species (ROS), which are small molecules that are highly reactive with proteins, nucleic acids, and lipids. ROS are potentially harmful to intracellular elements and their formation triggers cellular sensors that can engage signaling pathways involved in gene transcription (such as nuclear factor κB (NF-κB). While the exact mechanism of action is unknown, LLLT has been shown to interact with cytochrome c oxidase in mitochondria to release nitric oxide, facilitating oxidative phosphorylation. This increases ATP production and stimulates downstream signals to produce antioxidants and growth factors for cellular repair and proliferation. As a result, LLLT has been shown to decrease pain and inflammation and promote wound healing and tissue repair.

### 2.4 Product Efficacy

LLLT is a non-invasive technique which has been examined for the prevention and treatment of radiotherapy-induced OM. Multiple randomized trials have shown a reduction in the rates of OM and pain with the use of LLLT [11-20]. A list of trials examining the impact of LLLT for OM prevention in patients with HNC is given in table 1.

Furthermore, a systematic review and meta-analysis of eleven randomized placebo-controlled trials of LLLT use during chemotherapy or radiation therapy in HNC patients was performed [21]. This found a relative risk for developing OM was significantly (p=0.02) reduced after LLLT compared with placebo. The number of days with OM grade 2 or worse was also significantly reduced after LLLT to 4.38 days less than placebo. Likewise, OM severity was reduced after LLLT compared with placebo. All studies in this meta-analysis recorded possible adverse effects of LLLT therapy, but there were no differences from treatment with placebo. Evidence from these small, randomized controlled trials shows a significant reduction in incidence and severity of OM for HNC patients.

Additionally, the Multinational Association of Supportive Care in Cancer and International Society of Oral Oncology (MASCC/ISOO) Clinical Practice Guidelines for Mucositis recommends in favor of LLLT for the prevention of OM in patients receiving high-dose chemotherapy for hematopoietic stem cell transplants with or without total body irradiation and a suggestion for LLLT in the prevention of OM in patients receiving RT for HNC [22]. No guideline was issued for patients receiving concurrent chemotherapy and radiation therapy for HNC due to lack of high-level evidence. The European Society for Medical Oncology (ESMO) clinical practice guidelines for the management of oral and gastrointestinal mucositis also advises the use of LLLT to reduce the incidence of oral mucositis and its associated pain, in patients receiving high-dose chemotherapy or chemoradiotherapy before hematopoietic stem cell transplant [23].

Table 1. LLLT trials for oral mucositis prevention

| Reference | Population | Methods | Treatment | Results | Comments |
|---|---|---|---|---|---|
| Antunes et al<br>Radiother Oncol 2013[11] | HNC<br>(n=94)<br>Brazil, 2007-2010 | Phase III,<br>randomized<br>placebo controlled<br>trial | Concurrent Chemoradiotherapy (1) Placebosep (2) LLLT daily prior to each RT fraction Chemo: cisplatin 100 mg/m² q3weeks RT: 70.2 Gy LLLT: InGaAIP, 660 nm, 100mW, 1-4J/cm² | Grade 3-4 mucositis (WHO): 40.5% vs. 6.4% Relative risk: 0.16 (0.05 - 0.5) | Improved QOL for pain, swallowing and difficulty with eating |
| Arora et al<br>Oral Surg Oral Med Oral<br>Pathol Oral Radiol Endod<br>2008[13] | Oral cancer (n=50) India, 2005-2006 | Phase III,<br>randomized<br>controlled trial | Radiation (1) Topical anesthetic, saline washesser (2) LLLT daily prior to RT RT: 66 Gy LLLT: He-Ne, 632.8 nm, 10mW, 1.8J/cm <sup>2</sup> | Grade 3-4 mucositis (EORTC/RTOG) 53.9% vs. 18.2% at 3 weeks (p=0.019) | Functional impairment Scale maximum score: Oral alimentation not possible: 31% vs. 0% |
| Bensadoun et al<br>Support Care Center<br>1999[14] | HNC<br>(n=30)<br>France, 1994-1998 | Phase III,<br>randomized<br>placebo controlled<br>trial | Radiation (1) Placebose; (2) LLLT prior to each RT fraction RT: 65 Gy LLLT: He-Ne, 632.8 nm, 60mW, 2J/cm² | Grade 3 mucositis (WHO): 35.2% vs. 7.6% (p<0.01) Severe pain: 23.8% vs. 1.9% (p<0.05) | |
| Gautam et al<br>Radiother Oncol 2012[16] | HNC<br>(n=221)<br>India, 2009-2011 | Phase III,<br>randomized<br>placebo controlled<br>trial | Concurrent Chemoradiotherapy (1) Sham treatments (2) LLLT 5x/week, prior to or following RT Chemo: cisplatin 100 mg/m² q3weeks RT: 66 Gy LLLT: He-Ne, 632.8 nm, 24mW, 3J/point | Grade ≥3 mucositis (EORTC/RTOG): 70% vs. 23.4% (p < 0.0001) | Pain scores plateaued after<br>week 4 in LLLT arm and<br>continued to increase in<br>placebo arm<br>Lower dysphagia in LLLT arm |
| Zanin et al<br>Photomed Laser Surg<br>2010[18] | HNC<br>(n=72)<br>Brazil | Phase III,<br>randomized<br>controlled trial | Concurrent Chemoradiotherapy (1) No treatment (1) (2) LLLT 2x/week, prior to or following RT Chemo: cisplatin (1) (2) mg/m² weekly RT: 1.8 Gy daily fractions LLLT: He-Ne, 660 nm, 30mW, 2J/cm² | Mucositis (NCI) significantly lower in LLLT group from week 1 to week 4 (p=0.001), but remained stable until week 7 (p=0.68) | LLLT delayed onset of oral mucositis |
| Lima et al,<br>Braz Dent J 2010[17] | HNC<br>(n=25)<br>Brazil, 2005 | Prospective, non-<br>randomized study | RT ± chemotherapy (1) Sucrose and aluminum hydroxide suspension (2) LLLT daily prior to each RT fraction Chemo: cisplatin 100mg/m² q3weeks RT: 40-70 Gy LLLT: 830 nm, 60 mW, 12.4J/cm² | Grade 3 mucositis (OTS Scale) OM 50% vs. 33% (p=0.06) | Significant decrease in pain with LLLT (p=0.036) |

HNC; head and neck cancer. LLLT; low-level laser therapy. RT; Radiation. Gy; Gray. InGaAIP; indium phosphide, gallium and aluminum diode. nm; nanometer. mW; milliwatts. J; Joules. WHO; World Health Organization. QOL; Quality of Life. He-Ne; Helium-Neon. EORTC; European Organisation for Research and Treatment of Cancer. RTOG; Radiation Therapy Oncology Group. NCI; National Cancer Institute.

### 2.5 Product Safety

Lasers used for LLLT are categorized as Class 3b. Class 3b lasers emit 5mW to 500mW lasers, with some emitting infrared light below 5mW. A class 3b laser may be hazardous under direct and specular viewing conditions, but is not a fire hazard. The patient and LLLT operator require use of protective eyewear. The LLLT system is equipped with a key switch and a safety interlock. The THOR® Laser system (THOR Photomedicine Ltd, Chesham, UK) that will be used to deliver LLLT in this protocol is an FDA-approved medical device (510(K) number K030226).

There has been no reported toxicity in any of the studies of LLLT for the prevention and/or management of oral mucositis. In the limited number of studies evaluating extraoral LLLT, there has similarly been no reported cutaneous or oral toxicity.

### 2.6 Rationale for the Study

Previous phase III trials conducted in other countries, primarily Brazil [11], France [14], and India [16], have shown a significant improvement in OM with LLLT. However, no U.S. trials have been reported. The rationale for this phase II trial is to validate the results from international trials in a U.S. cohort of patients. Therefore, our goal is to evaluate the efficacy of LLLT in reducing treatment related toxicities including OM, pain, xerostomia, dysgeusia, and dysphagia and improving OM-related QOL in patients undergoing radiation with chemotherapy for HNC. To accomplish our goal, we propose a prospective, single-arm, phase II trial with the aim of improving health-care quality and reducing the incidence of treatment-related toxicity as compared to historical controls and a matched pair of control patients from our own institution.

# 3.0 Selection and Withdrawal of Subjects

### 3.1 Study Design

This is a phase II prospective, single-arm, open label trial testing the efficacy of LLLT in prevention of oral mucositis for HNC patients treated with chemoradiotherapy. Primary endpoints are the incidence of severe (assessed separately as CTCAE v. 4.0 grade 3-5 or WHO grade 3-4) OM in patients receiving a cumulative radiation dose of at least 5000 cGy. Secondary endpoints include the time onset to severe OM, mean cumulative radiation dose at the time of OM, duration of OM, the incidence of pain, dysphagia, xerostomia, dysgeusia, trismus, radiodermatitis, and QOL.

All toxicities will be graded by NCI CTCAE v. 4.0. In addition, oral mucositis will also be graded by WHO mucositis grading scale. Dysphagia will also be graded by a dietary assessment. Trismus will be assessed by measurements of the interincisal distance. QOL will be measured by the FACT-H&N assessment.

Previous studies (detailed in Section 2.2, Table 1) indicate that approximately 40% of patients will experience severe OM with radiation and concurrent chemotherapy. The hypothesis in this trial is that the addition of LLLT to this treatment regimen will decrease the rate of severe acute OM to 20%. We plan to enroll 50 patients at our institution in 12 months after the trial opens.

#### 3.2 Patient Selection

#### **Inclusion Criteria:**

- 1. Willing and able to understand and sign informed consent form approved by the HRPO.
- 2. Males or females greater than or equal to 18 years old.
- 3. Biopsy-proven HNC including cancers of the nasopharynx, oropharynx, larynx, hypopharynx, or HNC of unknown primary origin amenable to therapy with radiation and concurrent chemotherapy.
- 4. Patients who are planned to receive definitive or adjuvant radiotherapy with concurrent platinum-based chemotherapy.
- 5. Patients whose clinical treatment plans include a continuous course of external beam radiotherapy by intensity-modulated radiation therapy (IMRT) and/or image-guided radiation therapy (IGRT), given as a cumulative dose of 5000 7000 cGy in single daily fractions of 180 200 cGy, combined with a concurrent course of weekly or tri-weekly cisplatin or carboplatin chemotherapy.
- 6. Karnofsky performance status score >60.
- 7. Female subjects of child-bearing potential must have a negative pregnancy test prior to enrollment

#### **Exclusion Criteria:**

- 1. Subject has evidence of current mucositis, mucosal ulceration, or unhealed surgical wounds from surgical resection or biopsy.
- 2. Prior radiation to the head and neck.
- 3. Patients with gross tumor involvement of the oral cavity or oral mucosa.
- 4. Subjects planned to receive altered fractionation radiotherapy or multiple fractions per day
- 5. Subject is using a pre-existing feeding tube for nutritional support at the time of study entry.
- 6. Women who are pregnant or breast-feeding.
- 7. Subject plans to receive concurrent chemotherapy, other than the regimens specified in the inclusion criteria.
- 8. Patients who have chronic immunosuppression or are on current immunosuppressive therapies.
- 9. Patients who have a contraindication to radiation therapy.
- 10. Patients enrolled on another investigational trial for oral mucositis prevention.
- 11. Life expectancy of less than 3 months.
- 12. Unable or unwilling to adhere to study-specified procedures.

### 3.3 Withdrawal of Subjects

Any subject, having previously provided informed consent to participate in the protocol, is free to withdraw from the study at any time for any reason without prejudice to their future medical care by the physician or at the study site. The Investigator may also withdraw the subject at any time in the interest of subject safety. The primary reason for withdrawal must be recorded.

Subject participation may be terminated prior to completion of the clinical study for any of the following reasons:

- 1. Unacceptable toxicity
- 2. Death
- 3. Lack of efficacy
- 4. Withdrawal by subject

- 5. Lost to follow-up
- 6. Non-compliance with study treatment
- 7. Study physician decision in the best interest of subject safety
- 8. Pregnancy
- 9. Major protocol deviation that can affect the safety or efficacy of study population
- 10. Study terminated
- 11. Other

### 4.0 Treatment Methods

#### 4.1 Radiation Treatment

Prior to treatment, all patients will provide informed written for radiation therapy as per existing institutional policy. All patients will undergo a computed tomography (CT) simulation for treatment planning. Radiation therapy will be delivered with an intensity modulated radiation therapy (IMRT) technique and/or image-guided radiation therapy (IGRT). The prescribed course of radiotherapy will not be altered based on this study. Radiotherapy will be delivered 5 days per week, Monday – Friday with one radiation treatment given per day. The planned cumulative dose of radiation will be determined by the treating physician and will range from 5000 – 7000 cGy in 180 - 200 cGy daily fractions over the course of 5-7 weeks. This treatment is not part of the research protocol.

### **4.1.1 Definition of Target Volumes:**

Target volumes will be outlined per institutional practice and not modified based on this protocol. Target volumes are defined as the following:

*Gross Tumor Volume (GTV)* represents the region judged to contain gross primary tumor or involved node(s) based on clinical and endoscopic examinations, CT scan, and, when applicable, other imaging techniques.

Clinical Target Volume (CTV) is defined as the GTV plus areas considered at risk for containing microscopic disease delineated by the treating physician. The CTV margins can be narrower when GTV is in the proximity of the spinal cord or critical normal tissues.

*Planning Target Volume (PTV)* represents an additional margin around the CTV to compensate for the variability of treatment set up and internal organ motion.

#### 4.1.2 Definition of Organs at Risk:

CT-based planning will be used to identify the target volumes and organs at risk (OARs). OARs will be contoured according to the DAHANCA, EORTC, GORTEC, HKNPCSG, NCIC CTG, NCRI, NRG Oncology, and TROG consensus guidelines [24] which are included in table 2 which is provided in appendix 11.3. The dose parameters given to OARs will be recorded (table 3). Dose limits to OARs will be determined by institutional practice and specific dose-constraints will not be required on this protocol. The following radiation doses will be recorded.

#### Table 3. Dose parameters to OARs to be recorded

| Brainstem | Maximum Dose |
|-----------|--------------|

| Spinal Cord | Maximum Dose | |
|-----------------------------|--------------|-------------------|
| Right Parotid | Mean Dose | V30 <sub>Gy</sub> |
| Left Parotid | Mean Dose | V30 <sub>Gy</sub> |
| Parotids (bilateral) | D20cc | |
| Submandibular Gland | Mean Dose | |
| <b>Extended Oral Cavity</b> | Maximum Dose | Mean Dose |
| Lips | Maximum Dose | Mean Dose |
| <b>Buccal Mucosa</b> | Maximum Dose | Mean Dose |
| Mandible | Maximum Dose | |
| Pharyngeal Constrictors | Mean Dose | |

# 4.2 Chemotherapy

Prior to treatment, all patients will provide informed written for chemotherapy as per existing institutional policy. The prescribed course of chemotherapy will be determined by the managing medical oncologist per institutional practices and will not be altered based on this study. The frequency and dose of chemotherapy will be recorded for each patient on the trial. This treatment is not part of the research protocol.

## 4.3 Low-Level Laser Therapy

Treatment will be administered on an outpatient basis. While there are no expected toxicities, potential adverse events will be monitored per Section 7 (Adverse Events and Safety Monitoring). No investigational agents or therapies for the prevention of oral mucositis other than those described in this protocol may be administered.

LLLT will be delivered with the THOR® Laser system (THOR Photomedicine Ltd, Chesham, UK). LLLT will begin on the first or second day of radiotherapy and be delivered three times per week (Monday, Wednesday, and Friday) until the completion of radiotherapy. A trained radiation oncology nurse or physician will deliver treatment. LLLT may be delivered either immediately prior to or after the patient's daily fraction of radiotherapy. Patients will be treated extra-orally with a THOR® LED

cluster for one minute along the cheek to treat the buccal mucosa on each side and intraorally for one minute to the tongue and soft palate. During each LLLT treatment session a thorough oral exam will be performed to identify any areas of mucositis. If the patient should develop intraoral lesions they will be targeted directly with the intraoral probe for one minute to each site of mucositis.

The laser settings to be used are as follows: frequency 2.5 Hz; wavelength 660 nm; and power 75 mW. The dose per anatomic site treated will be 4.5 J/cm<sup>2</sup>.

The extra-oral probe will be cleaned before and after each use. Prior to each use, the intraoral probe will be covered with a protective dental sleeve. Patients and laser operator will wear THOR® laser safety glasses for the duration of laser therapy.

Treatment dates and sites will be recorded for each patient on the LLLT Treatment Record Form given in the appendix (appendix 11.4). Compliance with therapy will be documented. For each treatment session, the dose will be set (timer on control unit) and the patient will be positioned comfortably a chair. The LLLT device will be for a minimum of 3 exposures:

- 1. Right cheek
- 2. Left cheek
- 3. Tongue/Soft palate

The treatment per site will take 60 seconds, for a minimum treatment time of three minutes. If any areas of mucositis are evident on examination at the time of LLLT treatment, each area will be targeted with an intraoral probe for an additional 60 seconds.

There will be no pre- or post-treatment measures/precautions.

### 4.4 Other treatments

Subjects that develop symptomatic mucositis will be managed as necessary according to standard standard of care hospital protocol for oral mucositis in addition to LLLT. This may include topical creams, pain medications, anesthetic mouth rinses, mouth coatings, and nutritional support with supplementation either by mouth or feeding tube, without the use of specific investigational, restricted agents. No standard treatment will be denied to a patient on this protocol.

# 5.0 Follow-up and Assessments

### 5.1 Follow up Schedule

A general history & physical by a radiation oncologist and/or medical oncologist must be done within 8 weeks prior to registration. Patients will be evaluated for protocol eligibility at the time of initial consultation. At the time of initial evaluation, baseline assessments will be performed. During the course of treatment, each patient will be seen by the supervising physician in clinic for an ontreatment evaluation at least once per week (or at an interval of once per five radiation treatments). Follow-up appointments will be scheduled for two weeks and three months after the completion of therapy.

| Screening | Baseline | Treatment Period | | Treatment Period | Follow-up |
|---|---|---|---|---|---|
| | | Assessments LLLT Dosing | | Period | |
| Day -1 to | Study Day 0 | Weekly | 3x/week | Two weeks | |
| Day -28 | | | concomitant with | | |
| | | Last day of | chemoradiation | Three months | |
| | | treatment | | | |

# **5.2** Follow-up Assessments

During each assessment, the following toxicities will be assessed: pain, OM, dysphagia, xerostomia, dysgeusia, dermatitis, trismus, and QOL.

Mouth pain and throat pain severity will be assessed weekly using a standard 0-10 scale. A record of the amount of analgesic medications required will be required at each visit.

A diet assessment will be performed at weekly on-treatment assessments as follows:

| | Diet Ass | essment | |
|---|---|---|---|
| Diet 1: | Diet 2: | Diet 3: | |
| What has the subject been able to eat within the past 24 | If the subject has been unable to eat Solid food, mark all the reason(s) why (mark all that apply) | | Based solely on how the mouth feels, what does the |
| hours (mark only one) | | | subject feel (s)he could try to<br>eat if (s)he did not have to<br>swallow (mark only one) |
| □Solids | □Nausea/Vomiting | □Oral discomfort | □Solids |
| □Liquids | □Loss of appetite | □Dry mouth | □Liquids |
| □Nothing by Mouth | ☐Throat discomfort | □No teeth | □Nothing by Mouth |
| | □Difficulty Swallowing | | |
| If <b>Solids</b> is marked above, | □Other | | |
| proceed to next section. | | | |
| | If <b><u>Liquids</u></b> or <b><u>Nothing by</u></b> If <b><u>Oral discomfort</u></b> is marked above, proceed to | | |
| Mouth is marked about | the next section. | | |
| continue to "Diet 2". | If <b>Oral discomfort</b> is NO | | |
| | proceed to "Diet 3". | | |

OM will be assessed using the NCI CTCAE version 4.0 [25] as follows:

| Adverse<br>Event | Grade | | | | |
|---|---|---|---|---|---|
| | 1 | 2 | 3 | 4 | 5 |
| Oral<br>Mucositis | Asymptomatic or mild symptoms; intervention not indicated | Moderate pain; not interfering with oral intake; modified diet indicated | Severe pain;<br>interfering<br>with oral<br>intake | Life-threatening<br>consequences;<br>urgent<br>intervention<br>indicated | Death |

OM will also be assessed using the World Health Organization (WHO) grading scale [26]

| DM will also be assessed using the world Health Organization (wHO) grading scale [26]: | |
|---|---|
| WHO Oral Mucositis Grade | |
| Grade 0 (None) | None |
| Grade 1 (Mild) | Oral soreness/erythema |
| Grade 2 (Moderate) | Oral soreness/erythema, ulcers, can tolerate solid foods |

| Grade 3 (Severe) | Oral soreness/erythema, ulcers, liquid diet only |
|---|---|
| Grade 4 (Life-threatening) | Oral alimentation is not possible |

Patient-reported OM outcomes will be assessed using the Oral Mucositis Daily Questionnaire (OMDQ) [27]

#### **Oral Mucositis Daily Questionnaire**

2. During the PAST 24 HOURS how much MOUTH AND THROAT SORENESS DID YOU HAVE? (Circle one number)

| 0 | 1 | 2 | 3 | 4 |
|---|---|---|---|---|
| No soreness | A little soreness | Moderate soreness | Quite a lot of | Extreme soreness |
| | | | soreness | |

3. During the PAST 24 HOURS how much did MOUTH AND THROAT SORENESS limit you in each of the following activities:

| | Not limited | Limited a little | Limited some | Limited a lot | Unable to do |
|---|---|---|---|---|---|
| a. Swallowing | 0 | 1 | 2 | 3 | 4 |
| b. Drinking | 0 | 1 | 2 | 3 | 4 |
| c. Eating | 0 | 1 | 2 | 3 | 4 |
| d. Talking | 0 | 1 | 2 | 3 | 4 |
| e. Sleeping | 0 | 1 | 2 | 3 | 4 |

4. On a scale of 0 to 10, how would you rate your OVERALL MOUTH AND THROAT SORENESS during the PAST 24 HOURS? (*Please circle the most appropriate number*)

| 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 |
|------|---|---|---|---|---|---|---|---|-------|----------|
| None | | | | | | | | | Worst | possible |

<sup>\*</sup>Questions 2 through 4 of OMDQ adapted from Elting et al, 2008 [27]

Dysphagia will be assessed using the NCI CTCAE version 4.0 [25] as follows:

| Adverse<br>Event | Grade | | | | |
|---|---|---|---|---|---|
| Event | 1 | 2 | 3 | 4 | 5 |
| Dysphagia | Symptomatic,<br>able to eat<br>regular diet | Symptomatic and altered eating/swallowing | Severely altered<br>eating/swallowing;<br>tube feeding or TPN<br>or hospitalization<br>indicated | Life-threatening<br>consequences;<br>urgent<br>intervention<br>indicated | Death |

Xerostomia will be assessed using the NCI CTCAE version 4.0 [25] as follows:

| Adverse<br>Event | Grade | | | | |
|---|---|---|---|---|---|
| | 1 | 2 | 3 | 4 | 5 |
| Dry Mouth | Symptomatic (e.g., dry or thick saliva) without significant dietary alteration; unstimulated saliva flow >0.2 ml/min | Moderate symptoms; oral intake alterations (e.g., copious water, other lubricants, diet limited to purees and/or soft, moist foods); unstimulated saliva 0.1 to 0.2 ml/min | Inability to<br>adequately<br>aliment orally;<br>tube feeding or<br>TPN indicated;<br>unstimulated<br>saliva | - | - |

Dysgeusia will be assessed using the NCI CTCAE version 4.0 [25] as follows:

| Adverse<br>Event | Grade | | | | |
|---|---|---|---|---|---|
| | 1 | 2 | 3 | 4 | 5 |
| Dysgeusia | Altered taste but no change in diet | Altered taste with change in diet (e.g., oral supplements); noxious or unpleasant taste; loss of taste | - | - | - |

Dermatitis will be assessed using the NCI CTCAE version 4.0 [25] as follows:

| Adverse<br>Event | Grade | | | | |
|---|---|---|---|---|---|
| Lvent | 1 | 2 | 3 | 4 | 5 |
| Dermatitis<br>radiation | Faint erythema<br>or dry<br>desquamation | Moderate to brisk<br>erythema; patchy<br>moist desquamation,<br>mostly confined to<br>skin folds and<br>creases; moderate<br>edema | Moist<br>desquamation in<br>areas other than<br>skin folds and<br>creases; bleeding<br>induced by<br>minor trauma or<br>abrasion | Life-threatening<br>consequences;<br>skin necrosis or<br>ulceration of full<br>thickness dermis;<br>spontaneous<br>bleeding from<br>involved site; skin<br>graft indicated | Death |

#### **Trismus**

The interincisal distance will be measured in millimeters at the patient's maximum comfortable extent of mouth opening. Measurements will be taken at baseline, the last day of treatment, two-week follow-up, and 3 month follow-up appointments.

### **Quality of Life**

QOL will be assessed at the time of enrollment prior to initiation of treatment, on the last day of treatment, and on the last day of study participation, 3 months after completion of radiation. This will be assessed using the Functional Assessment of Cancer Therapy: General (FACT-G) version 4 (Appendix 11.7).

QOL as related to head and neck cancer will be assessed at each follow-up appointment using the FACT – H&N version 4 (Appendix 11.8).

### **6.0 Statistical Considerations**

### **6.1 Primary Endpoints:**

- The incidence of severe (WHO grade 3-4) oral mucositis in patients treated to a cumulative radiation dose of at least 5000 cGy.
- The incidence of severe (CTCAE v. 4.0 grade 3-5) oral mucositis in patients treated to a cumulative radiation dose of at least 5000 cGy.

### **6.2** Secondary Endpoints:

• Time to onset of severe (CTCAE v. 4.0 grade 3-4) oral mucositis following the initiation of radiotherapy.

- Mean cumulative radiation dose at time of onset of severe (CTCAE v. 4.0 grade 3-4) oral mucositis.
- Duration of oral mucositis.
- The incidence of pain.
- The incidence of dysphagia (CTCAE v. 4.0 and via diet assessment).
- The incidence of xerostomia (CTCAE v. 4.0).
- The incidence of dysgeusia (CTCAE v. 4.0).
- The incidence of trismus (Measurement of interincisal distance).
- The incidence of radiodermatitis (CTCAE v. 4.0).
- Evaluation of OM-related QOL (via FACT-H&N score).
- Incidence of any grade oral mucositis in patients treated to a cumulative radiation dose of at least 5000 cGy.

## **6.3** Exploratory Endpoints:

- Proportion of patients with severe (CTCAE v. 4.0 grade 3-4) oral mucositis by 5000 and 7000 cGy.
- Proportion of patients with severe (CTCAE v. 4.0 grade 3-4) oral mucositis by schedule of chemotherapy given (weekly versus Q 3 weeks).
- Time to reach planned dose of radiation therapy.
- Amount of narcotic analgesia use during treatment.
- Assessments of breaks in treatment defined as one of the following:
  - o Missing at least 1 chemotherapy treatment;
  - o Dose reduction in planned cisplatin administration; OR
  - o 3 consecutive days of no RT secondary to mucositis.
- Proportion of patients who require feeding tube placement during treatment (excluding patients who received a prophylactic feeding tube prior to the initiation of therapy).
- Percent change in body weight during the course of treatment.

### 6.4 Sample Size

Previous studies (detailed in Section 2.2, Table 1) indicate that approximately 40% of patients will experience severe OM with radiation and concurrent chemotherapy. The hypothesis in this trial is that the addition of LLLT to this treatment regimen will decrease the rate of severe acute OM to 20%. A sample size of 45 yields 90% power to detect a difference of 0.20 using an exact one-sided binomial test with a Type I error of 0.05. A total of 50 patients are required to ensure that there are at least 45 compliant with the treatment schedule. All patients should be enrolled in 12 months after the trial opens. We plan to enroll 50 patients at our institution.

# 6.5 Analysis

#### Primary endpoint

If 12 or fewer out of the 45 evaluable severe OM events occur, we will reject the null hypothesis that the occurrence of severe OM is 0.4 with the addition of LLLT therapy. Point and 90% confidence intervals (using Wilson's method) will also be estimated to describe the primary endpoint.

### Secondary endpoints

Descriptive statistics (point and exact 90% confidence interval estimates from the resultant Kaplan-Meier curve) will be generated for the time-to-severe OM and duration of severe OM endpoints. Point and 90% confidence intervals (using Wilson's method) will also be estimated to describe the binary endpoints. Continuous endpoints will be described by 90% confidence intervals using the t-distribution.

### **Exploratory endpoints**

Similar descriptive analyses as described in the above paragraph will be used for the binary, time-to-event and continuous endpoints.

### 6.6 Evaluation of Toxicity

All registered patients will be evaluated for toxicity probably related to the treatment. There have been no reported toxicities directly attributed to intraoral or extraoral LLLT. No systemic toxicities (e.g fever, nausea, fatigue) are anticipated or have been reported in association with oral LLLT. No specific toxicity is expected attributable to LLLT due to the addition of LLLT in patients receiving radiation with concurrent chemotherapy. Toxicity data will be collected at least weekly during the course of treatment to ensure the validity of this claim.

## **6.7** Specific Toxic Outcomes

No toxicities or dose-limiting toxicities have been reported in association with LLLT in the biomedical literature. Specifically with respect to LLLT for the prevention and/or management of oral mucositis, no toxicities or DLTs have been reported. Any toxicities arising would be anticipated to be localized to the exposed tissues. These would include undesignated skin/mucosal changes, such as localized skin erythema, mucosal swelling (not typically associated with mucositis) or unanticipated sensory changes. Of note, oral mucositis may develop despite LLLT and will not be considered a treatment-related toxicity.

We will closely monitor the following outcomes: grade 3 oral dysesthesia (burning/tingling sensation in the distribution exposed to LLLT), grade 3 or 4 oral mucosal swelling not attributable to mucositis (GI Disorders, other, specify), Grade 3 erythema and/or pain of the skin (in the distribution exposed to LLLT), visual loss, blurred vision, retinal tear or detachment, uveitis, or other eye disorders. If 2 or more patients out of the first 10 (or fewer) treated in the phase II portion of the study develop a grade III (using the CTCAE guidelines) or higher toxicity in any of these categories that are probably or definitely related to the LLLT treatment received within the first 2 weeks after the completion of treatment, we would recommend revisiting the study for safety reasons. Adjudication is necessary to ensure that we judge this study based on adverse events that are specific to LLLT therapy and not any other therapy that the patient happens to receive. We will continue to monitor these specific toxic outcomes throughout the course of the trial, in a sliding window fashion.

#### 6.8 Other toxic outcomes

Data on other toxic side effects (excluding those detailed in the previous paragraph) that patients may experience will also be collected. We have chosen a safety threshold of 0.25 to monitor other toxic side effects. We would recommend reconsidering the phase II portion of the study for safety reasons if there were X many occurrences of grade 3 or higher toxicity (using the CTCAE guidelines) among the first N (or fewer) patients treated, as it would result in an upper confidence limit greater than 0.25:

| N | X | p | UCL |
|----|---|-------|-------|
| 8 | 1 | 0.125 | 0.255 |
| 13 | 2 | 0.154 | 0.256 |
| 18 | 3 | 0.167 | 0.253 |
| 22 | 4 | 0.181 | 0.261 |
| 27 | 5 | 0.185 | 0.256 |
| 32 | 6 | 0.188 | 0.252 |
| 36 | 7 | 0.194 | 0.256 |
| 41 | 8 | 0.185 | 0.252 |

In the above table, N = the number of patients treated; X = the cumulative number of patients with a grade 3 or higher toxicity currently observed; p = the observed toxicity rate; and UCL = the exact 1-sided upper 80% confidence limit for p, using Wilson's method without a continuity correction. After treating 41 patients, the potential toxicity risk of this regimen should be well defined, and thereafter the possible need for termination of the study based on toxicity should be minimal.

### 6.9 Expected accrual rate, accrual duration, and study duration

Our anticipated accrual rate at our center is 50 patients per year. Thus, it should take approximately 1 year to accrue the maximum 50 patients needed for the data analysis. Allowing for 2 weeks of follow-up to obtain the primary endpoint on the last patient enrolled and 4 months to assemble, analyze and interpret the data the total study duration is projected to be at most 1.5 years.

# 7.0 Adverse Events and Safety Monitoring

least 3 months following the last LLLT treatment.

There have been no reported toxicities directly attributed to oral LLLT for the prevention/management of mucositis. Any toxicity would be expected to be localized to the region exposed (e.g. erythema of the skin, hyperalgesia). We do not anticipate treatment-related toxicity. LLLT has never been demonstrated to exacerbate or potentiate mucositis. Regardless, subjects will be followed carefully for any possible toxicity. Adverse event (AE) monitoring and reporting is a routine part of every clinical trial. These will be followed per Univ. of Pittsburgh requirements.

# 7.1 Reporting of Serious Treatment Emergent Adverse Events

An adverse event for the purposes of this protocol is the appearance of (or worsening of any pre-existing) undesirable sign(s), symptom(s), or medical condition(s) occurring after signing the informed consent even if the event is not considered to be related to the study drug(s). Please refer to the adverse event section of the protocol for the protocol-specific definitions of study drug and study treatment.

The descriptions and grading scales found in the revised NCI CTCAE version 4.0 will be utilized for AE reporting. All appropriate treatment areas should have access to a copy of the CTCAE version 4.0. A copy of the CTCAE version 4.0 can be downloaded from the CTEP web site <a href="http://ctep.cancer.gov/protocolDevelopment/electronic\_applications/ctc.htm">http://ctep.cancer.gov/protocolDevelopment/electronic\_applications/ctc.htm</a>. If CTCAE grading does not exist for an adverse event, the severity of mild, moderate, severe, and life-threatening, or grades 1 - 4, will be used. Adverse event monitoring should be continued for at

• 'Expectedness': AEs can be 'Unexpected' or 'Expected' for expedited reporting purposes only.

#### • **Attribution** of the AE:

- Definite The AE *is clearly related* to the study treatment.
- Probable The AE *is likely related* to the study treatment.
- Possible The AE *may be related* to the study treatment.
- Unlikely The AE *is doubtfully related* to the study treatment.
- Unrelated The AE *is clearly NOT related* to the study treatment.

Adverse events (but not serious adverse events) occurring before starting study treatment but after signing the informed consent form will be recorded as part of the medical history or current medical condition. Abnormal laboratory values or test results constitute adverse events only if they induce clinical signs or symptoms, are considered clinically significant or require therapy (e.g., any hematologic abnormality that requires transfusion or cytokine treatment); and should be recorded on the Adverse Events Case Report Form (CRF) under the signs, symptoms or diagnosis associated with them. In addition, isolated abnormal laboratory values that are considered clinically significant (e.g., cause study discontinuation or constitutes in and of itself a Serious Adverse Event) should be recorded on the Adverse Events CRF. SAEs occurring after signing the Informed Consent are recorded on the Adverse Event CRF.

#### 7.2 Adverse Event Characteristics

The occurrence of adverse events should be sought by non-directive questioning of the patient at each visit during the study. Adverse events also may be detected when they are volunteered by the patient during or between visits or through physical examination, laboratory test, or other assessments. As far as possible, each adverse event should be evaluated to determine:

- 1. The severity grade (CTCAE grade 1-4)
- 2. Its relationship to each study treatment (suspected/not suspected)
- 3. Its duration (start and end dates or if continuing at final exam)
- 4. Action taken (no action taken/temporarily interrupted; study treatment permanently discontinued due to this adverse event; concomitant medication taken; non-drug therapy given; hospitalization/prolonged hospitalization)
- 5. Whether it is serious, where a serious adverse event (SAE) is defined as one which:
  - Is fatal or life-threatening
  - Results in persistent or significant disability/incapacity
  - Constitutes a congenital anomaly/birth defect
  - Requires inpatient hospitalization or prolongation of existing hospitalization, unless hospitalization is for:
  - Routine treatment or monitoring of the studied indication, not associated with any deterioration in condition (specify what this includes)
  - Elective or pre-planned treatment for a pre-existing condition that is unrelated to the indication under study and has not worsened since signing the informed consent
  - Treatment on an emergency outpatient basis for an event not fulfilling any of the definitions of a SAE given above and not resulting in hospital admission
  - Social reasons and respite care in the absence of any deterioration in the patient's general condition
  - Is medically significant, i.e., defined as an event that jeopardizes the patient or may require medical or surgical intervention to prevent one of the outcomes listed above

Unlike routine safety assessments, SAEs are monitored continuously and have special reporting requirements; see protocol section on Serious Adverse Event reporting.

All adverse events should be treated appropriately. Once an adverse event is detected, it should be followed until its resolution, an assessment should be made at each visit (or more frequently, if necessary) of any changes in its severity, its suspected relationship to the study treatment, any of the interventions required to treat it, and its outcome.

Information about all serious adverse events will be collected and recorded. A serious adverse event is an undesirable sign, symptom or medical condition which:

- is fatal or life-threatening
- results in persistent or significant disability/incapacity
- constitutes a congenital anomaly/birth defect
- requires inpatient hospitalization or prolongation of existing hospitalization, unless hospitalization is for:
  - routine treatment or monitoring of the studied indication, not associated with any deterioration in condition (specify what this includes)
  - elective or pre-planned treatment for a pre-existing condition that is unrelated to the indication under study and has not worsened since the start of study drug
  - treatment on an emergency outpatient basis for an event not fulfilling any of the definitions of a SAE given above and not resulting in hospital admission
  - social reasons and respite care in the absence of any deterioration in the patient's general condition
- is medically significant, i.e., defined as an event that jeopardizes the patient or may require medical or surgical intervention to prevent one of the outcomes listed above

Events **not** considered to be serious adverse events are hospitalizations for the routine treatment or monitoring of the studied indication, not associated with any deterioration in condition.

- Sores in the mouth and throat that are likely to interfere with swallowing
- Temporary hair loss (of the face/chin/neck)
- Tanning, redness, or blistering or peeling of skin in treatment area
- Loss of teeth, or cavities in teeth, if strict dental care is not followed
- Hardness and tightness of the skin and muscles of the head and neck
- Dryness of the mouth or altered taste that may be permanent
- Loss of appetite
- Weight loss which may necessitate the placement of a temporary feeding tube
- Nausea and/or vomiting
- Weakness
- Hearing loss, ringing of the ears
- Numbness of the fingers and toes
- Lower blood counts with risk of infection or bleeding
- Anemia
- Loss of taste
- Muscle cramps
- Loss of coordination
- Involuntary movement
- Restlessness
- Treatment, which was elective or pre-planned, for a pre-existing condition that did not worsen

• Treatment on an emergency, outpatient basis for an event **not** fulfilling any of the definitions of serious given above and **not** resulting in hospital admission.

### 7.3 HRPO Adverse Event reporting

Investigators must report the following to the Univ. of Pittsburgh Human Research Protection Office:

- Internal Adverse Events that are (i) Unexpected, (ii) Related or Possibly Related to the Research Intervention, and (iii) serious or otherwise suggests that the research places the subject or others at a greater risk of harm (including physical, psychological, economic or social harm) than was previously known or recognized.
- External Adverse Events that are (i) Unexpected; (ii) Related to the Research Intervention and (iii) Serious or otherwise suggests that the research places subjects or others at greater risk than was previously recognized.

Adverse Events that meet the University HRPO's reporting requirements must be reported to the HRPO office as follows:

- Internal Adverse Events which are unexpected, fatal or life-threatening, and related or possibly Related to the Research Intervention must be reported to the HRPO within 24 hours of learning of the event. (Note: It is recognized that the information available during this 24 hour period may not be sufficient to permit accurate completion of the required adverse event reporting forms. However, the HRPO should, at a minimum, be notified of the fatal or life-threatening internal adverse event during this time frame, with subsequent followup submission of a more detailed written report.)
- All other internal Adverse Events will be reported to the HRPO within 10 working days of the investigator learning of the event.
- External Adverse Events which are Unexpected, Serious AND suggest that the research places subjects or others at greater risk than was previously recognized, and Related to the Research Intervention will be reported to the HRPO within 30 working days of their receipt by the University/UPMC investigator.

### 7.4 Data Safety Monitoring

A data safety monitoring board will meet monthly to evaluate toxicity for this trial.

During these meetings the investigators will discuss:

- Safety of protocol participants (adverse events and reporting)
- Validity and integrity of the data (data completeness on case report forms and complete source documentation)
- Enrollment rate relative to expectation of target accrual, (eligible and ineligible participants)
- Retention of participants, adherence to the protocol and protocol violations
- Protocol amendments

Patients/adverse events will be discussed at these monthly disease center meetings. Unexpected serious adverse events will be reported to the HRPO and radiation oncology data safety monitoring board (DSMB), and minutes of the monthly disease center meetings will be reviewed at the DSMB meetings

Any clinically significant or unexpected disease or condition that is found during the course of this study, will be immediately evaluated by the Principal Investigator and appropriate medical staff and then it will be determined how to proceed with the study/ study treatment.

#### 7.5 Ethics

The study will be performed in accordance with ethical principles that have their origin in the Declaration of Helsinki and are consistent with ICH/Good Clinical Practice, applicable regulatory requirements.

The final study protocol, including the final version of the Written Informed Consent Form, must be approved in writing by the Univ. of Pittsburgh HRPO.

The principal investigator is responsible for informing the Univ. of Pittsburgh HRPO of any amendments to the protocol. The protocol must be re-approved by the HRPO annually. Progress reports and notifications of serious, unexpected adverse events or drug reactions will be provided to the HRPO.

The principal investigator will ensure that the subject is given full and adequate oral and written information about the nature, purpose, possible risk and benefit of the study. Subjects must also be notified that they are free to discontinue from the study at any time. The subject should be given the opportunity to ask questions and allowed time to consider the information provided. In accordance with the Health Information Portability and Accountability Act (HIPAA), the Written Informed Consent Form must include a subject authorization to release medical information to any agency, or Institutional Review Board access to subject's medical information that includes all hospital records relevant to the study, including subjects' medical history.

The principal investigator must store the original, signed Written Informed Consent Form. A copy of the signed Written Informed Consent Form must be given to the subject.

# 8.0 Registration Procedures

#### 8.1 General Guidelines

Eligible patients will be entered on the study at UPMC Shadyside Department of Radiation Oncology, by the Study Coordinator.

At the time of registration:

- Patients must have signed an informed consent form prior to registration.
- Confirm that all required pre-study requirements are completed as per the study calendar.
- Collect demographic information on the patient including age, gender, smoking history, alcohol history, tumor stage, histology, prior therapy.

### **8.2** Registration Process

To register a patient, the following documents should be completed and faxed or e-mailed to the Study Coordinator:

• Signed patient consent form

### 9.0 Protocol Conduct and Guidelines

### 9.1 Protocol amendments, or changes in study conduct

Any change or addition (excluding administrative) to this protocol requires a written protocol amendment that must be reviewed and approved. Amendments significantly affecting the safety of subjects, the scope of the investigation or the scientific quality of the study require additional approval by the HRPO.

If an immediate change to the protocol is felt to be necessary by the investigator and is implemented for safety reasons the HRPO must be informed immediately. Amendments affecting only administrative aspects of the study do not require formal protocol amendments or HRPO approval but the HRPO must be kept informed of such administrative changes.

#### 9.2 Publication of results

The results of this study will be presented in abstract form in an international medical conference forum and published in a peer-reviewed journal.

#### 9.3 Ethics and Good Clinical Practice

This study must be carried out in compliance with the protocol and the principles of Good Clinical Practice, as described in:

- ICH Harmonized Tripartite Guidelines for Good Clinical Practice 1996. Directive 91/507/EEC, The Rules Governing Medicinal Products in the European Community.
- US 21 Code of Federal Regulations dealing with clinical studies (including parts 50 and 56 concerning informed consent and IRB regulations).
- Declaration of Helsinki and amendments, concerning medical research in humans (Recommendations Guiding Physicians in Biomedical Research Involving Human Subjects).

The investigator agrees to adhere to the instructions and procedures described in it and thereby to adhere to the principles of Good Clinical Practice that it conforms to.

### 9.4 Institutional Review Board/Independent Ethics Committee

Before implementing this study, the protocol, the proposed informed consent form and other information to subjects, must be reviewed by a properly constituted Institutional Review Board/Independent Ethics Committee/Research Ethics Board (IRB/IEC/REB).

#### 9.5 Informed consent

The investigator must explain to each subject (or legally authorized representative) the nature of the study, its purpose, the procedures involved, the expected duration, the potential risks and benefits involved and any discomfort it may entail. Each subject must be informed that participation in the study is voluntary and that he/she may withdraw from the study at any time and that withdrawal of consent will not affect his/her subsequent medical treatment or relationship with the treating physician.

This informed consent should be given by means of a standard written statement, written in non-technical language. The subject should read and consider the statement before signing and dating it,

and should be given a copy of the signed document. If the subject cannot read or sign the documents, oral presentation may be made or signature given by the subject's legally appointed representative, if witnessed by a person not involved in the study, mentioning that the patient could not read or sign the documents. No patient can enter the study before his/her informed consent has been obtained.

The informed consent form is considered to be part of the protocol, and must be submitted by the investigator with it for IRB/IEC/REB approval.

### 9.6 Declaration of Helsinki

The investigator will conduct the trial in accordance with the principles of the Declaration of Helsinki. Copies of the Declaration of Helsinki and amendments will be provided upon request or can be accessed via the website of the World Medical Association at http://www.wma.net/e/policy/17-c e.html.

# 10.0 References

- 1. Pfister, D.G., et al., *Head and Neck Cancers, Version 1.2015.* J Natl Compr Canc Netw, 2015. **13**(7): p. 847-56.
- 2. Trotti, A., et al., *Mucositis incidence, severity and associated outcomes in patients with head and neck cancer receiving radiotherapy with or without chemotherapy: a systematic literature review.* Radiother Oncol, 2003. **66**(3): p. 253-62.
- 3. Cheng, K.K., et al., Severe oral mucositis associated with cancer therapy: impact on oral functional status and quality of life. Support Care Cancer, 2010. **18**(11): p. 1477-85.
- 4. Groome, P.A., et al., Compromised local control due to treatment interruptions and late treatment breaks in early glottic cancer: Population-based outcomes study supporting need for intensified treatment schedules. Int J Radiat Oncol Biol Phys, 2006. **64**(4): p. 1002-12.
- 5. Elting, L.S., et al., *Risk, outcomes, and costs of radiation-induced oral mucositis among patients with head-and-neck malignancies.* Int J Radiat Oncol Biol Phys, 2007. **68**(4): p. 1110-20.
- 6. Huang, Y.Y., et al., *Biphasic dose response in low level light therapy an update.* Dose Response, 2011. **9**(4): p. 602-18.
- 7. Kim, W.S. and R.G. Calderhead, *Is light-emitting diode phototherapy (LED-LLLT) really effective?* Laser Ther, 2011. **20**(3): p. 205-15.
- 8. Sutherland, J.C., *Biological effects of polychromatic light.* Photochem Photobiol, 2002. **76**(2): p. 164-70.
- 9. Karu, T., *Laser biostimulation: a photobiological phenomenon.* J Photochem Photobiol B, 1989. **3**(4): p. 638-40.
- 10. Karu, T.I. and S.F. Kolyakov, *Exact action spectra for cellular responses relevant to phototherapy.* Photomed Laser Surg, 2005. **23**(4): p. 355-61.
- 11. Antunes, H.S., et al., *Phase III trial of low-level laser therapy to prevent oral mucositis in head and neck cancer patients treated with concurrent chemoradiation.* Radiother Oncol, 2013. **109**(2): p. 297-302.
- 12. Arun Maiya, G., M.S. Sagar, and D. Fernandes, *Effect of low level helium-neon (He-Ne) laser therapy in the prevention & treatment of radiation induced mucositis in head & neck cancer patients.* Indian J Med Res, 2006. **124**(4): p. 399-402.
- 13. Arora, H., et al., *Efficacy of He-Ne Laser in the prevention and treatment of radiotherapy-induced oral mucositis in oral cancer patients.* Oral Surg Oral Med Oral Pathol Oral Radiol Endod, 2008. **105**(2): p. 180-6, 186 e1.
- 14. Bensadoun, R.J., et al., Low-energy He/Ne laser in the prevention of radiation-induced mucositis. A multicenter phase III randomized study in patients with head and neck cancer. Support Care Cancer, 1999. **7**(4): p. 244-52.
- 15. Gautam, A.P., et al., Low level laser therapy against radiation induced oral mucositis in elderly head and neck cancer patients-a randomized placebo controlled trial. J Photochem Photobiol B, 2015. **144**: p. 51-6.
- 16. Gautam, A.P., et al., Low level laser therapy for concurrent chemoradiotherapy induced oral mucositis in head and neck cancer patients a triple blinded randomized controlled trial. Radiother Oncol, 2012. **104**(3): p. 349-54.
- 17. Lima, A.G., et al., *Efficacy of low-level laser therapy and aluminum hydroxide in patients with chemotherapy and radiotherapy-induced oral mucositis.* Braz Dent J, 2010. **21**(3): p. 186-92.
- 18. Zanin, T., et al., *Use of 660-nm diode laser in the prevention and treatment of human oral mucositis induced by radiotherapy and chemotherapy.* Photomed Laser Surg, 2010. **28**(2): p. 233-7.

- 19. Carvalho, P.A., et al., Evaluation of low-level laser therapy in the prevention and treatment of radiation-induced mucositis: a double-blind randomized study in head and neck cancer patients. Oral Oncol, 2011. **47**(12): p. 1176-81.
- 20. Oton-Leite, A.F., et al., *Effect of intraoral low-level laser therapy on quality of life of patients with head and neck cancer undergoing radiotherapy.* Head Neck, 2012. **34**(3): p. 398-404.
- 21. Bjordal, J.M., et al., *A systematic review with meta-analysis of the effect of low-level laser therapy (LLLT) in cancer therapy-induced oral mucositis.* Support Care Cancer, 2011. **19**(8): p. 1069-77.
- 22. Lalla, R.V., et al., *MASCC/ISOO clinical practice guidelines for the management of mucositis secondary to cancer therapy.* Cancer, 2014. **120**(10): p. 1453-61.
- 23. Peterson, D.E., et al., *Management of oral and gastrointestinal mucositis: ESMO Clinical Practice Guidelines.* Ann Oncol, 2011. **22 Suppl 6**: p. vi78-84.
- 24. Brouwer, C.L., et al., *CT-based delineation of organs at risk in the head and neck region:*DAHANCA, EORTC, GORTEC, HKNPCSG, NCIC CTG, NCRI, NRG Oncology and TROG consensus guidelines. Radiother Oncol, 2015. **117**(1): p. 83-90.
- 25. Institute, N.C., *Common Terminology Criteria for Adverse Events v4.0* in *NIH publication # 09-7473*, N. NCI, DHHS. , Editor.
- 26. Organization, W.H., *WHO handbook for reporting results of cancer treatment*. 1979: Geneva: World Health Organization.
- 27. Elting, L.S., et al., *Patient-reported measurements of oral mucositis in head and neck cancer patients treated with radiotherapy with or without chemotherapy: demonstration of increased frequency, severity, resistance to palliation, and impact on quality of life.* Cancer, 2008. **113**(10): p. 2704-13.